CLINICAL TRIAL: NCT03068364
Title: Additive Value of Biological and Electrocardiographic Biomarkers for Risk Stratification in Hypertension
Brief Title: Biological and Electrocardiographic Biomarkers for Risk Stratification in Hypertension.
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0151
Record Dates: First submitted 2017-02-27; First posted 2017-03-01 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
Keywords: Mortality; Hypertension; Left ventricular hypertrophy; NT-proBNP; ECG; Transthoracic echocardiography
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Risk stratification of hypertensive patients includes assessment of traditional cardiovascular risk factors and subclinical target organ damages particularly left ventricular hypertrophy (LVH).

LVH may routinely screened by transthoracic echocardiography by measuring the left ventricular mass (LVM).

However, transthoracic echocardiography suffers from several pitfalls: poor reproducibility, technical limitations and unavailability at a first evaluation by general practitioners.

Other biomarkers may be particularly helpful in hypertension risk stratification. The amplitude of the R wave in aVL lead is a simple validated ECG parameters of LVH and a strong predictor of cardiovascular events and mortality.

Plasma N-terminal pro Brain Natriuretic Peptide (NT-proBNP) is also strongly related to LVM and is an independent predictor of all-cause mortality in hypertension.

The main objective of our study is to determine the additive prognostic value of R wave in aVL and NT proBNP on all-cause and cardiovascular mortality.

Secondary objectives are to determine the addition prognostic value of NT-proBNP and R wave in aVL combined in comparison to each marker taken into account

This study will include 1600 patients who had a work-up of their hypertension in the Cardiology Department of Croix-Rousse Hospital (Hospices Civils de Lyon, Lyon, France) from January 1997 to January 2014.

Their data will be collected in an Access database; their vital status will be obtained by the INSEE unit CépiDC.

ELIGIBILITY:
* Inclusion Criteria:

  * >18 years old
  * men or women
  * questionnaire completion and physical exam during their first stay in the Cardiology Department of from January 1997 to January 2014.
* Exclusion Criteria:

  * Patients refusal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients, who had a work-up of their hypertension in the Cardiology Department of Croix-Rousse Hospital (Hospices Civils de Lyon, Lyon, France) from January 1997 to January 2014.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
All- cause and cardiovascular mortality in hypertension | an average of 7 years
  All-Cause and cardiovascular mortality will be obtained from the INSERM unit CépiDC.
  Vital status was obtained in July 2016

SECONDARY OUTCOMES:
All-cause and cardiovascular deaths | an average of 7 years
  All-cause and cardiovascular deaths in the study population will be obtained from the INSERM unit CépiDC.
  Vital status was obtained in July 2016

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LANTELME, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse, Lyon, France